CLINICAL TRIAL: NCT06902948
Title: Effectiveness of a Standardized Stroke Upper Limb Rehabilitation Program with Shortened Fugl-Meyer Assessment Stratification: a Randomized Controlled Trial
Brief Title: Effectiveness of a Standardized Stroke Upper Limb Rehabilitation Program with Shortened Fugl-Meyer Assessment Stratification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sally Hiu Lam Wong (Other Government)
Responsible Party: Sponsor-Investigator, Sally Hiu Lam Wong, Advanced Practice Physiotherapist, Tai Po Hospital
Organization: Tai Po Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CREC2022.343-T
Record Dates: First submitted 2025-03-16; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: Shortened Fugl-Meyer Assessment; stroke rehabilitation; upper limb
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standardized upper limb rehabilitation program (Experimental): A new stroke upper limb rehabilitation program was designed. Participants were classified into 3 categories based on their level of upper limb impairment reflected by the baseline S-FM score (severe 0-4, moderate 5-8, mild 9-12). Upper limb training was provided according to the standardized treatment choices preset with expert opinions
  Interventions: Other: upper limb function training
- Conventional upper limb training (Active Comparator): Treatments were prescribed based on the corporate stroke rehabilitation protocol of Hong Kong Hospital Authority. The protocol allowed variations in clinical practice and ultimate decision about a particular clinical treatment depended on each individual patient's condition and clinical judgment of individual therapists.
  Interventions: Other: upper limb function training

INTERVENTIONS:
Other: upper limb function training — Intervention selection included stretching and mobilization exercise, strengthening exercise, electrical stimulation, acupuncture, functional or task specific training and mirror therapy.

SUMMARY:
The objective of the study was to investigate the effectiveness of a standardized stroke upper limb rehabilitation program with stratification using Shortened Fugl-Meyer Assessment (S-FM). The standardized program was compared with conventional training based on the hospital protocol.

ELIGIBILITY:
Inclusion Criteria:

* first stroke, able to attend gym training and give written consent

Exclusion Criteria:

* unstable medical condition, any musculoskeletal conditions or other diseases restricted upper limb training, unfit mental state and unable to follow command

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Shortened Fugl-Meyer Assessment (S-FM) | From enrollment to the end of treatment up to 6 weeks
  S-FM consisted of six items examining upper extremity movements (shoulder elevation, shoulder flexion 90° to 180°, elbow extension, elbow 90° pronation/supination, elbow 90° wrist flexion/extension and grasp, adduct thumb). Each item was scored with an ordinal scale of 0 (unable to perform), 1 (partially performed) and 2 (fully performed). The total score was 12.
Functional Test for the Hemiplegic Upper Extremity (FTHUE) | From enrollment to the end of treatment up to 6 weeks
  FTHUE consisted of 18 activities examining upper extremity function. Seven levels with 1-3 activities in each level in a hierarchy sequence of difficulty were adopted.

SECONDARY OUTCOMES:
Modified Barthel Index (MBI) | From enrollment to the end of treatment up to 6 weeks
  MBI consisted of 11 items examining ADL including self-care, continence and locomotion. A modified scoring system with 5 codes (unable to perform task, attempts task but unsafe, moderate help required, minimal help required and fully independent) was adopted for each item, giving a total score from 0 to 100 (0= fully dependent, 100= fully independent).

CONTACTS AND LOCATIONS:
Locations (1):
- Tai Po Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years
Access Criteria: Researchers who are working on similar study topic with approved independent review can contact for IPD and supporting information sharing. A proposal that describes planned analyses and signed data sharing agreement have to be submitted to the corresponding author for review.

REFERENCES:
- [Background] McDonnell MN, Hillier SL, Esterman AJ. Standardizing the approach to evidence-based upper limb rehabilitation after stroke. Top Stroke Rehabil. 2013 Sep-Oct;20(5):432-40. doi: 10.1310/tsr2005-432. PMID 24091285
- [Background] Garcia-Vega J, Gregory G, Lind CRP, Singer BJ. Development of a consensus approach to upper limb rehabilitation early post stroke amongst a cohort of Western Australian therapists. N Z J Physiother 2016;44(3):133-147
- [Background] Hirayama K, Takebayashi T, Takahashi K. Factors Influencing Decision-Making for Poststroke Paretic Upper Limb Treatment: A Survey of Japanese Physical and Occupational Therapists. Occup Ther Int. 2024 Oct 7;2024:1854449. doi: 10.1155/2024/1854449. eCollection 2024. PMID 39403110
- [Background] Hsieh YW, Hsueh IP, Chou YT, Sheu CF, Hsieh CL, Kwakkel G. Development and validation of a short form of the Fugl-Meyer motor scale in patients with stroke. Stroke. 2007 Nov;38(11):3052-4. doi: 10.1161/STROKEAHA.107.490730. Epub 2007 Oct 4. PMID 17916763
- [Derived] Lam Wong SH, Tung Chim TH, Ho Chung BP, On Lau TF. Effectiveness of a standardised stroke upper extremity rehabilitation program with shortened Fugl-Meyer assessment stratification: A randomised controlled trial. Hong Kong Physiother J. 2025 Dec;45(2):157-167. doi: 10.1142/S1013702525500131. Epub 2025 Nov 25. PMID 41477567